CLINICAL TRIAL: NCT04948632
Title: A Medico-Economic Evaluation of a Telehealth Platform for Elective Outpatient Surgeries: a Trial Study
Brief Title: Optimization of Outpatient Surgery at the CHUM Using the LeoMed Telecare Platform
Acronym: MEET-OS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: HEC Montreal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21.110
Record Dates: First submitted 2021-06-28; First posted 2021-07-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Surgery--Complications; Patient Satisfaction; Quality of Life
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, controlled study comparing, in patients undergoing outpatient surgery at the CHUM, a group of patients benefiting from optimized support and follow-up using the LeoMed telecare platform (Group A) with a group benefiting from the current standard of care (Group B).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete LeoMed application (Active Comparator): LeoMed application with integrated artificial intelligence
  Interventions: Other: Complete LeoMed application
- Basic LeoMed application (Placebo Comparator): LeoMed application without artificial intelligence
  Interventions: Other: Basic LeoMed application

INTERVENTIONS:
Other: Complete LeoMed application — Access to the complete LeoMed application on the participant's smartphone. The day before surgery, participants will receive notifications encouraging them to use the platform to help prepare for their surgery. Safety instructions will also be sent. Postoperatively, notifications will be sent to the participants every day during the first 4 days and on the 7th day. These notifications will direct them to online forms that aim to assess their condition. On the 15th and 30th postoperative day, the platform will send a follow-up form. The platform will collect this information and classify it for appropriate management of their condition.
  Arms: Complete LeoMed application
Other: Basic LeoMed application — Access to a partial version of the LeoMed application on the patient's smartphone during a visit to the preoperative clinic. Before surgery, participants will receive a phone call to be summoned to the hospital and to remind them of the safety instructions. Postoperatively, their follow-up will not be standardized and will vary depending on their surgeon. On the 15th and 30th postoperative day, the platform will send a follow-up form. In the event of an emergency, they will receive the contact details of the CHUM Health Infoline to ensure the continuity of their care.
  Arms: Basic LeoMed application

SUMMARY:
The main objective of this study is to carry out a medico-economic evaluation of a new platform for outpatient surgical care, by comparing the effectiveness and utility of the deployment of this trajectory on patients and the health system to a control group.

DETAILED DESCRIPTION:
Outpatient surgery allows the patient to leave the hospital on the day of their surgery and thus avoid complete hospitalization. There are many advantages to this practice. Patients can remain in the comfort of their own home with the support of their family caregivers and the healthcare system can avoid incurring additional hospital costs and redirect these savings to other critical needs. However, despite the advantages of outpatient surgery, the tools and measures currently in place to supervise the preparation before the operation and the follow-up after the operation are suboptimal.

Following surgery, adverse events such as moderate to severe pain, nausea/vomiting, infection and bleeding from the operative site are very rarely sought out and detected by healthcare facilities. However, these are the main causes of readmissions or emergency consultations for patients.

In order to optimize the care offer, the anesthesiology department, the innovation and artificial intelligence center of the CHUM as well as the Quebec telecare platform LeoMed have joined forces in order to offer, through a health application, follow-up and personalized support for patients undergoing outpatient surgery.

The investigators believe that the integration of this platform in the course of care will allow early diagnosis of the main postoperative complications and therefore, prevent calls to the Health-Info line, emergency room returns, as well as readmissions or unscheduled postoperative consultations.

A patient-as-partner approach has been chosen in the initial phase, where 12 patients having had an outpatient surgery less than 6 months ago, will be recruited to test the platform. Another 12 patients, scheduled to undergo an outpatient surgery, will test the optimized support and follow up application. Their feedback will help to correct and/or improve the platform, if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old undergoing elective outpatient surgery under general or regional anesthesia
* Internet access for the patient or their caregiver from home
* Written, oral and spoken comprehension of French or English

Exclusion Criteria:

* Patient's or caregiver's inability to learn and use digital technologies
* Conversion of outpatient to inpatient hospitalization on the day of surgery
* Patient's refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness analysis of the LeoMed® telecare platform | 1 month after the surgery
  The cost-effectiveness of the telecare platform deployment will be evaluated by the assessment of direct costs. These costs include unanticipated cancellations of the surgery on the day of surgery, calls at the CHUM local health info line, calls at the Quebec health info line (811), visits to the emergency department, unplanned readmissions or medical visits (family physician or outpatient clinic) for a problem related to the procedure.

SECONDARY OUTCOMES:
Cost-utility analysis of the LeoMed® telecare platform | Change between baseline (pre-operative) and 1 month postoperative
  The cost-utility analysis of the telecare platform will be evaluated with the improvement of patient's quality of life. The EQ-5D-5L-VAS will be used to assess quality of life. It is a valid questionnaire including five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Patient satisfaction with care services will also be assessed.
  Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to /extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level for each of the five dimensions.
  The VAS portion of the questionnaire EQ-5D-5L-VAS is a scale where patients are asked to indicate their overall health on the day that the questionnaire is completed, 0 = the worst health you can imagine and 100 = the best health you can imagine.
Patient satisfaction | 1 month after the surgery
  Patient satisfaction with care services and the telecare platform will also be assessed and compared between the two groups using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Robin, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Robin F, Roy M, Kuftedjian A, Perret L, Lavoie F, Castonguay A, Pomey MP, Zaouter C, Pare G. A Medicoeconomic Evaluation of a Telehealth Platform for Elective Outpatient Surgeries: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Apr 24;12:e44006. doi: 10.2196/44006. PMID 37093634